CLINICAL TRIAL: NCT03890055
Title: Clinical Study of First-line Treatment of Small Cell Lung Cancer (SCLC) With Anlotinib Hydrochloride in in Combination With EC/EP
Brief Title: Clinical Study of First-line Treatment of Small Cell Lung Cancer (SCLC) With Anlotinib Hydrochloride
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chifeng Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B19267BT
Record Dates: First submitted 2019-03-24; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical trial group (Experimental): （Carboplatin/cisplatin + etoposide）+ （Anlotinib Hydrochloride 12 mg/day ，Each cycle was defined as 2 weeks on-treatment fol- lowed by 1 week off-treatment）, after 4-6 cycles of treatment, the treatment was continued with anlotinib until disease progression.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Best supportive care
  Other Names: Focusv

SUMMARY:
This study was designed to investigate the efficacy and side effects of combining erlotinib with classical EC/EP chemotherapy regimens.

DETAILED DESCRIPTION:
Lung cancer is a common malignant tumor that poses a serious threat to human health. Small cell lung cancer accounts for about 20% of lung cancer. Precision medicine has recently been perfectly interpreted in many tumor types, but the treatment of small cell lung cancer is still bleak. The EC/EP regimen is the most classic chemotherapy regimen for small cell lung cancer with good results but is prone to drug resistance. In 2018, with the development of immunotargeting therapy, small molecule multi-target anti-angi drugs, PARP inhibitors, new chemotherapy drugs, etc., the treatment of small cell lung cancer has ushered in a new dawn. As a kind of highly selective multi-target anti-angiogenic TKI drugs,Anlotinib Hydrochloride is a kind of 1.1 innovative drugs with independent intellectual property rights in China, mainly acting on VEGFR, PDGFR, FGFR and c-Kit. The latest ALTER1202 study confirms that anlotinib is significantly improved for PSC and ORR in SCLC patients who have previously received at least 2-line chemotherapy. OS data is not yet mature, but the benefits of the anlotinib group were observed. The adverse effects of anlotinib were consistent with expectations, no new adverse events were found, and safety was tolerated. Nowadays, the effective combination of traditional chemical therapy with molecular targeting and immunotherapy is the future development direction of lung cancer treatment. Therefore, this topic is designed to combine the efficacy of safety and safety with the treatment of anlotinib with the classic EC/EP chemotherapy regimen. Expected to get longer PFS and OS for patient benefit.

ELIGIBILITY:
Inclusion Criteria:

1. patients 18-75 years of age.
2. A metastatic or recurrent advanced SCLC confirmed by histology or cytology and did not receive any other treatment;
3. a measurable disease
4. an Eastern Cooperative Oncology Group PS of 0-1;
5. an estimated survival duration of >6 months;

Exclusion Criteria:

1. Have used erlotinib or other anti-vascular targeted drugs (eg, Endo, bevacizumab, etc.)2. Patients who have been treated with chemotherapy or radiotherapy for previous tumors.3.Have appeared or merged with other tumors within 5 years.4.Patients with no measurable lesions; 5.any severe and uncontrolled disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
PFS | nine months
  progression-free survival

SECONDARY OUTCOMES:
OS | 12 months
  overall survival
ORR | 12 months
  Objective Response Rate
DCR | 12 months
  disease control rate
safety assessed by Adverse reactions | 12 months
  Adverse reactions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Han JY, Kim HY, Lim KY, Han JH, Lee YJ, Kwak MH, Kim HJ, Yun T, Kim HT, Lee JS. A phase II study of sunitinib in patients with relapsed or refractory small cell lung cancer. Lung Cancer. 2013 Feb;79(2):137-42. doi: 10.1016/j.lungcan.2012.09.019. Epub 2012 Nov 20. PMID 23182663
- See also: National Institutes of Heaith — https://www.nih.gov/